CLINICAL TRIAL: NCT02864784
Title: A Prospective, Multicenter, Randomized, Placebo-Controlled, Two-armed, Double-blind Pilot Study to Evaluate the Safety, Tolerability and Efficacy of ACC vs. Placebo for the Treatment of Subjects With Castrate Resistant Prostate Cancer With Bone Metastasis
Brief Title: Investigating the Safety, Tolerability and Efficacy of Amorphous Calcium Carbonate (ACC) on the Treatment of Subjects With CRPC
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Budget
Sponsor: Amorphical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMCS-ONCO-PR-001-CTIL
Record Dates: First submitted 2016-08-02; First posted 2016-08-12 (Estimated); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Castrate Resistant Prostate Cancer With Bone Metastasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amorphous calcium carbonate (Experimental): Subjects in this arm of the study will receive ACC tablets, containing 200 mg elemental calcium in addition to the standard treatment with ZA or Denosumab (4 mg once every 4 weeks for ZA and 120mg (1.7ml injection) every 4 weeks for Denosumab)
  Interventions: Drug: Amorphous calcium carbonate
- Placebo (Placebo Comparator): Subjects in this arm of the study will receive Placebo tablets in addition to standard treatment with ZA or Denosumab (4 mg once every 4 weeks for ZA and 120mg (1.7ml injection) every 4 weeks for Denosumab)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Amorphous calcium carbonate — Subjects in this arm of the study will receive standard treatment with ZA or Denosumab (4 mg once every 4 weeks for ZA and 120mg (1.7ml injection) every 4 weeks for Denosumab) as well as AMOR-1 tablets, containing 200 mg elemental calcium per tablet, individually titrated up to the maximum level which does not induce grade 2 hypercalcemia.
  Other Names: ACC
  Arms: Amorphous calcium carbonate
Other: Placebo — microcrystalline cellulose
  Arms: Placebo

SUMMARY:
Studies objectives:

To evaluate the safety, tolerability and efficacy of ACC given in combination with ZA or with Denosumab as compared to placebo given with ZA or with Denosumab as outline below:

* Safety and Tolerability:
* Adverse events (AEs) and serious AEs
* Safety laboratory measurements
* Hypercalcemic and hypercalciuric episodes
* Treatment withdrawal due to AEs and overall

Efficacy:

* Skeletal Related Events (SREs)
* Measurable and evaluable disease progression
* Progression Free Survival (PFS)
* Pain assessment via the VAS scale

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 year
2. Histologic proof of Castrate Resistant Prostate Cancer with Bone Metastasis
3. Systemic steroids are only allowed if needed for hormonal therapy
4. Previous radiation therapy must have been completed more than four weeks prior to enrollment into this study, unless subjects are under radiotherapy as a rescue therapy. Subjects must have recovered from all side effects.
5. The last dose of chemotherapy must have been completed at least four weeks prior to enrollment into this study, and subjects must have recovered from all side effects.
6. Subjects must have a performance status of 0-2 by the ECOG Scale.
7. Subjects must have pretreatment (obtained < 7 days prior to treatment) granulocyte count of > 2,000/μL, platelet count of > 100,000/μL, WBC > 3,000/μL, hemoglobin ≥ 10.0 g/dL, serum creatinine < 1.5 mg/dL, bilirubin < 1.5 mg/dL, and ALT/AST not more than 3x the upper limit of normal (or not more than 5x if the elevation is due to liver metastases).
8. Subjects must be normo-calcemic upon study entry.
9. Subjects must be Vitamin D sufficient upon study entry, which is defined as 25(OH)D serum level >20 ng/mL (50 nmol/L) according to a document composed by the Food and Nutrition Board of the Institute of Medicine, USA. If the subject is Vitamin D insufficient or deficient, then a loading dose of Vitamin D3 will be administered as follows:

   * If the serum 25(OH)D level is 12-20 ng/mL (30-50 nmol/L) then a loading oral dose of 50,000 IU of Vitamin D3 should be administered twice with 3-5 days in between the doses.
   * If the serum 25(OH)D level is ≤ 12 ng/mL (30 nmol/L), then a loading oral dose of 50,000 IU of Vitamin D3 will be administered three times with 3-5 days in between the doses. Serum 25(OH)D levels will be checked 1-2 weeks following the last loading.
10. Regardless of Vitamin D levels, all subjects will receive a daily maintenance dose of 1000 IU Vitamin D3, which should be taken in the morning with breakfast.
11. Estimated life expectancy of > 3 months.
12. Subjects must be accessible for follow-up.
13. Written informed consent will be obtained.

Exclusion Criteria:

1. Concurrent treatment with acute anticancer therapy
2. Hormonal and corticosteroid therapies for Skeletal Related Events are not allowed
3. Sarcoidosis
4. Hypercalcemia
5. Hypophosphatemia
6. Hypoparathyroidism/Hyperparathyroidism
7. Major surgery within 4 weeks of anticipated inception of AMOR-1therapy
8. Serious intercurrent infections or non-malignant medical illnesses that are uncontrolled or whose control may be jeopardized by the complications of therapy
9. Psychiatric disorders rendering subjects incapable of complying with the requirements of the protocol
10. Any illness or condition deemed by the investigator to contra-indicate treatment with AMOR-1 or ZA or Denosumab
11. Hypersensitivity to ZA or Denosumab or Abiraterone acetate or Enzalutamide, or to any bisphosphonates or to any of the following excipients: Mannitol and Sodium citrate.
12. Active cancer treatment except hormonal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Changes in the number of Skeletal Related Events (SREs) | Bone scan will take place at baseline and week 12

SECONDARY OUTCOMES:
Time from randomization to onset of first SRE. | Bone scan will be made on baseline and week 12
Proportion of subjects (%) with SREs. | Bone scan will take place at baseline and week 12
Proportion of subjects (%) with evidence of measureable and evaluable disease progression or SREs. | Bone scan will take place at baseline and week 12
Progression Free Survival (PFS). | CT or MRI will be assessed on screening and week 12
Number of subjects that are receiving radiation as a rescue treatment | An assessment will take place at week 2,4,6,8,10,12 16,20 and 24
Frequency and incidence of treatment emergent adverse events (TEAEs) | Safety assessment will take place at week 2,4,6,8,10,12 16,20 and 24
Frequency and incidence of serious treatment emergent adverse events (TEAEs). | Safety assessment will take place at weeks 2,4,6,8,10,12 16,20 and 24
Proportion of subjects (%) with hypercalcemic DLTs. | Safety assessment will be made at weeks 2,4,6,8,10,12 16,20 and 24
Proportion of subjects (%) with any DLTs. | Safety assessment will take place at weeks 2,4,6,8,10,12 16,20 and 24
Number of hypercalciuric events. | Urine calcium levels will be examined by urine tests, taking place at weeks 4,8,12,16,20 and 24

CONTACTS AND LOCATIONS:
Locations (1):
- Soroka Medical Center, Beersheba, Israel

IPD SHARING:
Plan to Share IPD: No